CLINICAL TRIAL: NCT05121025
Title: Pathogen-microbiome Interaction in Human Response and Disease-outcome During Infection and Colonization With Helicobacter Pylori
Brief Title: Pathogen-microbiome Interaction During Helicobacter Pylori Infection
Acronym: PREDICTHP
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Mohamed Tarek Badr, Principal Investigator, University Hospital Freiburg
Other Study IDs: 21/1552
Record Dates: First submitted 2021-10-25; First posted 2021-11-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Metagenomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Helicobacter pylori patients: Patients with gastric biposies which was positive for Helicobacter pylori in culture
  Interventions: Diagnostic Test: Analysis of gut microbiome and immune signatures
- Helicobacter pylori asymptomatic carriers: Healthy controls who are positive for Helicobacter pylori antigen in stool and have no symptoms of gastritis
  Interventions: Diagnostic Test: Analysis of gut microbiome and immune signatures
- Healthy controls: Healthy controls who are negative for Helicobacter pylori antigen in stool and have no symptoms of gastritis
  Interventions: Diagnostic Test: Analysis of gut microbiome and immune signatures

INTERVENTIONS:
Diagnostic Test: Analysis of gut microbiome and immune signatures — The investigators will analyse the microbiome composition (16S rDNA-sequencing and metagenomics), microbiome activity (RNA-sequencing of stool bacteria and metabolite sampling) and immune cell activity (leukocyte RNA-sequencing) of all study groups.

SUMMARY:
Helicobacter pylori affects the gut microbiome in ways that are only partially understood. In which patients H. pylori causes severe disease and in whom it merely colonizes, possibly even with beneficial effects, is not understood. The investigators are pursuing the hypothesis that changes in the gut microbiome that can be easily measured in stool have such predictive value.

DETAILED DESCRIPTION:
Helicobacter pylori colonizes the stomach of about half of the world's population, including about 20-30% of adults in Germany. In some cases, this colonization can lead to chronic inflammation of the gastric mucosa, which can lead to various serious diseases such as ulcer disease and gastric cancer. It has been reported several times in the literature that Helicobacter pylori infection negatively affects the human intestinal flora and can lead to microbial imbalance (dysbiosis). Recent studies, mostly from mouse models, reveal new roles and interactions of the microbiome: host immune response may influence bacterial activity; bacterial metabolites may determine microbiome functions. Differences in the microbiome were also found between Helicobacter pylori-infected patients and were associated with treatment success. On the other hand, beneficial microbial symbiosis may prevent intestinal inflammation. The reasons for these differences in the microbiome of Helicobacter pylori-infected patients, which may also contribute to treatment failure, remain to be investigated. Therefore, this project aims to investigate how Helicobacter pylori affects the bacteria and fungi of the human gastrointestinal microbiome and how the suspected microbial imbalance may influence treatment success. In this project, The investigators aim to answer the question of how these newly discovered mechanisms alter the course of human H. pylori infection. The investigators will analyze H. pylori itself in colonized patients and asymptomatic individuals (whole genome sequencing), determine the immune response of the carrier (RNA expression in lymphocytes), and composition of the gut microbiome (DNA sequencing) and activity (RNA expression in the bacteria/fungi and identification of metabolites). Using bioinformatics approaches, particularly machine learning, The investigators will determine the parameters that predict disease progression and eradication success. The results will provide important decision support for H. pylori-infected patients.

ELIGIBILITY:
Inclusion Criteria:

Patients: -

* Male and female patients aged ≥ 18 years.
* Specimens from patients undergoing tissue sampling, stool, and blood to rule out Helicobacter pylori infection
* Written informed consent from patients.

Volunteer subjects: -

* Male and female (non-pregnant) volunteers between the ages of 18-65 years.
* Written informed consent from volunteers.
* No acute medical conditions
* No regular medication use, and no antibiotic use in the last 4 weeks.

Exclusion Criteria:

Patients: -

* Minor patients
* Patients not capable of giving consent
* Samples without sufficient residual material after standard diagnostic procedures
* Samples from patients who have not given consent for testing

Volunteer subjects: -

* Subjects not capable of giving consent
* Subjects with acute illnesses
* Subjects older than 65 or younger than 18 years of age.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of full age who are capable of giving consent and from whom gastric biopsies, stool, and whole blood/serum will be obtained for diagnostic purposes (to exclude Helicobacter pylori infection), irrespective of the clinical picture. The indication for specimen collection is made by the treating clinical physician independent of the study. Patients should be informed about the study by the treating clinician concurrently with being informed about the risk of biopsy collection. Healthy volunteers will be invited to donate stool and blood for H. pylori diagnostics.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori microbiome and immune signatures | 12-18 Months
  The diversity of the gut microbial species of patients and controls as well as transcriptomic signatures of blood immune cells will be assessed and compared to conclude specisifc signatures that are associated with the disease and carrier status. These signatures will be analyzed to identify specific bacterial and immune biomarkers that can be used as a screening tool for Helicobacter pylori infection.

SECONDARY OUTCOMES:
Helicobacter pylori eradication control | 12-24 Months
  Patients with positive gastric biopsy for Helicobacter pylori will be assessed for successful eradication after treatment, and the eradication success will be compared with the patients' microbial signatures to identify specific gut microbial signatures that are associated with treatment outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Microbiology and Hygiene, Freiburg im Breisgau, Baden-Wurttemberg, Germany